CLINICAL TRIAL: NCT03602222
Title: Increasing Provider Competence for Treating Stress-related Mental Health Conditions in Low Resource Settings
Brief Title: An LGBT-Competency Program for Mental Health Professionals in Romania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Corina Lelutiu-Weinberger, Assistant Professor, Rutgers University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RutgersU
Record Dates: First submitted 2018-06-15; First posted 2018-07-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Stigma, Social; Gays; Lesbians; Bisexuals; Gender Dysphoria
Keywords: LGBT mental health; provider training in LGBT-affirmative clinical practice
MeSH Terms: conditions — Social Stigma; Homosexuality; Homosexuality, Female; Bisexuality; Gender Dysphoria

STUDY DESIGN:
Intervention Model Description: 120 MHPs will be randomized to receive the training either in-person or mobile on the web, concomitantly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person training LGBT mental health (Active Comparator): In-person training LGBT mental health: Participants randomized to the in-person condition will receive training in LGBT-affirmative mental health counseling face-to-face.
  Interventions: Behavioral: In-person training LGBT mental health
- Mobile training LGBT mental health (Experimental): Mobile training LGBT mental health: Participants randomized to the mobile training condition will receive training in LGBT-affirmative mental health counseling while on the web.
  Interventions: Behavioral: Mobile web training LGBT mental health

INTERVENTIONS:
Behavioral: Mobile web training LGBT mental health — Mobile web training LGBT mental health: Half of the participants were randomly assigned to receive the training in LGBT mental health in a the mobile fashion (on the web).
  Arms: Mobile training LGBT mental health
Behavioral: In-person training LGBT mental health — In-person training LGBT mental health: Half of the participants were randomly assigned to receive the training in LGBT mental health in-person.
  Arms: In-person training LGBT mental health

SUMMARY:
Lesbian, gay, bisexual and transgender individuals (LGBTI) present increased morbidity compared to the general population, which is attributed to healthcare discrimination and lack of LGBT-specific expertise, especially in high-stigma countries. Motivated by fear, Romanian LGBTI conceal their identities and report significantly more barriers to healthcare access than heterosexuals. Poor mental health, specifically anxiety and depression, is elevated for Romanian LGBTI, and associated with poor physical health (e.g., HIV risk, alcohol abuse.) However, LGBT-competent mental health professionals (MHPs) are nearly non-existent in Romania, and thus the negative impact of homophobia on mental health cannot be ameliorated. Given that a pilot of an in-person LGBT-affirmative MHP training recently tested in Romania showed significant receptivity and increased competence among MHPs, this training is ripe for testing its feasibility and efficacy in creating significant change via mobile delivery, in a randomized controlled trial (RCT). Proving the efficacy of this first mobile training and supervision model has high potential for cost-effective and expeditious boundless dissemination. Aim 1 will test the relative feasibility and efficacy of the mHealth MHP training by conducting an RCT comparing a mobile training (MT) of MHP LGBT-competency program (n=60) to the equivalent in-person training (IPT) (n=60) recently piloted. Both programs' content and structure will be identical (2-day trainings and two boosters 6 months apart). At baseline, 4, 8, and 12 months, all MHPs' LGBT-related attitudes, knowledge of LGBT health needs and clinical practice, and LGBT caseload will be assessed in a mobile fashion. In Aim 2 will test the efficacy of a companion mHealth supervision and consultation program in maintaining LGBT competency and enhancing LGBT-friendly practice. Half of the MHPs in each group will receive mHealth supervision and expert consultation program, consisting of monthly 2-hour virtual group meetings to discuss case studies, in order to determine the added benefit of mobile supervision. At the end of the study, 10 MHPs will provide interview-based program feedback. In Aim 3, the investigators will build mHealth research capacity among MHPs by demonstrating how to integrate mobile data collection tools in clinical practice to monitor client progress for personalized treatment plans.

DETAILED DESCRIPTION:
Participants and Procedures. Partner Consortium. The PI has strategically chosen four types of partners in order to maximize the sustainability of our training. The study team's multidisciplinarity will increase the potential for reach across domains that are pivotal in changing the landscape of mental health for LGBTI in Romania. First, the team partnered with a multi-service provider, the Romanian Association against AIDS (ARAS), a non-governmental not-for-profit organization founded in 1992 to support the health of hidden and vulnerable groups including LGBTI. ARAS intends to expand the depth and breadth of its LGBT-competency in mental health. Second, the team has received the essential support of academics (Hyperion University and Professors Călugaru and Dumitriu), which are forefront agents for social change. Third, individual MHPs in private practice who are connected with key associations have signed on as liaisons to their affiliated organizations (e.g., Bellanima Center for Psychotherapy and Psychiatry) to facilitate training participation. Fourth, the team continues its fruitful collaboration with their technical developer, Data Center Solutions (DCS), who built the mobile platform on which the team delivered live therapy for DMDN, collected real-time mental health and behavioral data, and disseminated sexual health materials. DCS is an expert in health systems information technology (medical e-learning; patient health-promotion), and will build our mHealth training platform.

Inclusion Criteria. 120 Romanian practicing MHPs (psychologists or psychiatrists) or MHPs in training will be eligible to participate.

Recruitment. The Partner Consortium will advertise the project via web-postings, listservs and eblasts to their national circles. Facebook ads were the most successful source of recruitment for DMDN. The team will thus be able to canvas all regions of Romania. Further, due to the pilot work, the team is maintaining contact with close to 100 MHPs from Bucharest (the capital), and other cities (e.g., Sibiu, Iasi, Cluj Napoca, Timisoara). While they will not be eligible to participate because they had exposure to the program, they will circulate, as indicated by their Letters of Support, future trainings among their circles of individual practice and professional affiliations (e.g., Romanian Collegiate of Psychologists, the Cognitive Behavioral Therapy Association of Romania).

Screening and Consent. Study ads will link to the Qualtrics electronic screener easily accessed from any mobile device. MHPs will take the 5-minute survey (Appendix 2) to determine eligibility, and be randomized to either the MT group or IPT group (based on age and geographical region). The study budgeted travel stipends for one-third of the MHPs, whom the team anticipate live outside Bucharest, such that travel costs will not impede their participation in IPT and to ensure that each group will include samples that are unbiased geographically. Notably, the pilot included non-Bucharest residents. Alternate training dates will be offered for those unable to attend the trainings. Group assignment, training dates, locations, and link to a Qualtrics baseline (BL) survey will be sent prior to the training. The BL contains the consent form with our contacts for questions. The team tested these procedures in the pilot, during which the PI answered study questions from MHPs via email.

Sixty MHPs will be randomized to receive a 2-day IPT in Bucharest, and 60 MHPs will be randomized to the equivalent 3-day MT, on a DCS-designed platform compatible with any mobile device, and with document-sharing and voice-conferencing capabilities. The didactic trainings will be interspersed with answering MHP's questions (voice or text).

Supervision and Consultation. After the first follow-up (4 months post training), half of the IPT MHPs and half of the MT MHPs (n=30 per group, total n=60) will receive 2-hour monthly mobile supervision using a forum format on our mobile platform for 8 months. DCS will design a group chat feature, similar to the one they devised for a previous pilot study. The live monthly supervision will occur on this platform after the 4-month and before the 12-month assessments. This system will provide MHPs with a fully automated and interactive mobile platform through which they will participate in supervision, as well as submit questions and receive answers for case consultation from the experts (Dr. Pachankis and DMDN intervention psychologists) within 48 hours. Further, MHPs will receive case studies through our mobile website, monthly, with response options asking them their best approach to helping the client (e.g., common LGBT stressor situations such as coming out, negotiating sexual safety, reducing isolation, or replacing health-depleting behaviors such as excessive drinking with healthy alternatives). Cases are fully discussed during supervision. At the end of the study, those who did not receive supervision will be given access to all the case studies and the mobile consultation site to achieve equity.

Boosters. We will hold two 2-hour IPT and MT boosters, respectively, 6 and 12 months post training, and provide an overview of LGBT-affirmative therapy principles, their incorporation into clinical practice, clarifications, and troubleshooting. Case studies will be included covering common issues raised by LGBTI.

Measures of MHP Attitudes, Knowledge, and Clinical Practice. The mixed-methods design involves qualitative interviews (n=10) and 30-min. self-administered internet-based quantitative surveys (n=120) by MHPs, the latter being administered at BL, and at 4, 8, and 12-month follow-ups. Surveys will be identical and assess, in a mobile fashion, changes in MHPs' LGBT attitudes, knowledge of LGBT health needs, clinical practice skills, and LGBT caseload.

Feasibility and Acceptability. Feasibility measures include data on session attendance. Acceptability measures include 5-min. session rating surveys (on mobile devices), and the 10 qualitative interviews.

Efficacy. MHPs will report their age, gender, specialization, years of clinical practice, and LGBT caseload. We will measure attitudes, knowledge and clinical skills; and the presence of explicit and implicit stigma and homophobia.

ELIGIBILITY:
Inclusion Criteria:

* Romanian practicing MHPs (psychologists or psychiatrists) or MHPs in training

Exclusion Criteria:

* All those who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in attitudes towards LGBT patients as assessed by the Attitudes Subscale of the Sexual Orientation Provider Competency Scale | Change in negative attitudes (mean scores) from baseline to each follow-up assessment point (4, 8, and 12 months post-training )
  The Attitudes Subscale of the Sexual Orientation Provider Competency Scale measures providers' negative attitudes towards LGBT clients. It consists of 10 items rated on a 5-point Likert scale ranging from 1, ''strongly disagree,'' to 5, ''strongly agree.'' A higher score indicates more negative attitudes.
Changes in knowledge for LGBT competent practice as assessed by the Knowledge Subscale of the Sexual Orientation Provider Competency Scale | Change in Knowledge (mean scores) from baseline to each follow-up assessment point (4, 8, and 12 months post-training )
  The Knowledge Subscale of the Sexual Orientation Provider Competency Scale measures providers' LGBT knowledge of issues that are specific to LGBT clients. It consists of 8 items rated on a 5-point Likert scale ranging from 1, ''strongly disagree,'' to 5, ''strongly agree.'' A higher score indicates more knowledge.
Changes in clinical skills as assessed by the Clinical Skills subscale of the Sexual Orientation Provider Competency Scale | Change in Clinical Skills (mean scores) from baseline to each follow-up assessment point (4, 8, and 12 months post-training )
  The Clinical Skills Subscale of the Sexual Orientation Provider Competency Scale measures providers' clinical skills in addressing LGBT mental health issues. It consists of 8 items rated on a 5-point Likert scale ranging from 1, ''strongly disagree,'' to 5, ''strongly agree.'' Item 7 was reverse-coded. A higher score indicates more clinical skills.
Changes in homophobic attitudes towards LGBT patients as assessed by the Modern Homonegativity Scale | Change in homophobic attitudes (mean scores) from baseline to each follow-up assessment point (4, 8, and 12 months post-training )
  The Modern Homonegativity Scale measures providers' homophobic attitudes towards LGBT individuals. It consists of 11 items rated on a 5-point Likert scale ranging from 1, ''strongly disagree,'' to 5, ''strongly agree.'' Items 5 and 8 were reverse-coded. A higher score indicates higher homophobic attitudes.
Changes in implicit bias attitudes towards homosexual (gay or lesbian) individuals as assessed by the Sexual Orientation Implicit Association Test (Sexual Orientation IAT) | Change in implicit bias (mean scores) from baseline to each follow-up assessment point (4, 8, and 12 months post-training )
  The Sexual Orientation IAT measures providers' implicit bias against homosexual (gay or lesbian) individuals. It consists of a reaction-time double categorization task in which participants are asked to categorize positive (e.g., "joyful") or negative (e.g., "disgusting") concepts and images of homosexual or heterosexual couples. Scores range between -1 and +1, with scores closed to 0 indicating impartial attitudes towards either group, scores closer to -1 indicating lower implicit bias towards homosexual individuals.

SECONDARY OUTCOMES:
LGBT client case load | Change (increase) in LGBT client case load (total number reported) from baseline to each follow-up assessment point (4, 8, and 12 months post-training )
  The number of LGBT clients a mental health professional has. Higher intervention impact is indicated by increases in LGBT client load at each follow-up assessment point post-training.
Intervention Feasibility measured by session attendance | Feasibility (session attendance) will be measured at baseline, and the two boosters at 6 months and 12 months post-baseline. An indicator of high feasibility includes 120 attendees for the training and two boosters.
  Feasibility measures include data on session attendance. These numbers should ideally be as close to 120 for the training sessions and booster sessions (6 and 12 months post training) as possible to indicate high intervention feasibility.
Intervention Acceptability measured by session rating surveys | The session ratings will take place at the end of the training. The training consisted of 2 days and it was held approximately two weeks after baseline.
  Acceptability measures include 5-minute session rating surveys of the quality of the training. It consists of 9 items rated on a 5-point Likert scale ranging from 1, ''strongly disagree,'' to 5, ''strongly agree.'' The higher the score is, the higher the acceptability.
Intervention Acceptability measured by qualitative interviews | The 10 qualitative interviews will take place at the end of the study (12 months post training).
  Acceptability measures include 10 phone qualitative interviews with randomly selected trainees. These cannot be quantified, but themes will be identified (e.g., concept clarity, content appropriateness, missing information) indicative of positive and negative aspects identified by interviewees, informing how acceptable the training was and what changes need to be made for future iterations of it.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Lelutiu-Weinberger, PhD, Study Director — Rutgers University
Locations (1):
- ARAS, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
All those interested should contact the PI who will then share relevant study information.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available August 2019, indefinitely.
Access Criteria: All interested parties should contact the PI.